CLINICAL TRIAL: NCT04978506
Title: Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Multiple Rising Oral Doses of BI 1569912 (Single-blind, Partially Randomized Within Dose Groups, Placebo-controlled, Parallel Group Design) With an Optional Posology (Uptitration) Part (Single-blind, Partially Randomized Within Dose Groups, Placebo-controlled, Parallel Group Design) in Healthy Male Subjects
Brief Title: A Study in Healthy Men to Test How Well Different Doses of BI 1569912 Are Tolerated
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1447-0002; 2021-001717-36 (EudraCT Number)
Record Dates: First submitted 2021-07-26; First posted 2021-07-27 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- BI 1569912 MRD: treatment group 1 (Experimental): Multiple rising dose (MRD) part
  Interventions: Drug: BI 1569912
- BI 1569912 POSO treatment group (Experimental): Posology part (optional)
  Interventions: Drug: BI 1569912
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- BI 1569912 MRD: treatment group 2 (Experimental): Multiple rising dose (MRD) part
  Interventions: Drug: BI 1569912
- BI 1569912 MRD: treatment group 3 (Experimental): Multiple rising dose (MRD) part
  Interventions: Drug: BI 1569912
- BI 1569912 MRD: treatment group 4 (Experimental): Multiple rising dose (MRD) part
  Interventions: Drug: BI 1569912
- BI 1569912 MRD: treatment group 5 (Experimental): Multiple rising dose (MRD) part
  Interventions: Drug: BI 1569912
- BI 1569912 MRD: treatment group 6 (Experimental): Multiple rising dose (MRD) part
  Interventions: Drug: BI 1569912
- BI 1569912 elderly treatment group (Experimental)
  Interventions: Drug: BI 1569912

INTERVENTIONS:
Drug: BI 1569912 — BI 1569912
  Arms: BI 1569912 MRD: treatment group 1; BI 1569912 MRD: treatment group 2; BI 1569912 MRD: treatment group 3; BI 1569912 MRD: treatment group 4; BI 1569912 MRD: treatment group 5; BI 1569912 MRD: treatment group 6; BI 1569912 POSO treatment group; BI 1569912 elderly treatment group
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The main objectives of this trial are to investigate (1) safety, tolerability, pharmacokinetics and pharmacodynamics following multiple rising doses of BI 1569912; (2) tolerability of BI 1569912 in an up-titrating dosing scheme.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (Blood pressure (BP), pulse rate (PR)), 12-lead electrocardiogram (ECG), and clinical laboratory tests
* MRD- and POSO-part: Age of 18 to 45 years (inclusive); ELDERLY-part: Age of 65 to 80 years (inclusive)
* Body mass index (BMI) of 18.5 to 29.9 kg/m2 (inclusive)
* Signed and dated written informed consent prior to admission to the study, in accordance with GCP and local legislation
* Male subjects who meet any of the following criteria from at least 30 days before the first administration of trial medication until 30 days after trial completion:

  * Use of adequate contraception, e.g. any of the following methods (of female partners) plus condom: implants, injectables, combined oral or vaginal contraceptives, intrauterine device
  * Sexually abstinent
  * Surgically sterilised (including hysterectomy of female partner)
  * Postmenopausal female partner, defined as at least 1 year of spontaneous amenorrhea (in questionable cases a blood sample with follicle stimulating hormone (FSH) above 40 U/L and estradiol below 30 ng/L is confirmatory)

Exclusion Criteria:

* Any finding in the medical examination (including BP, PR or ECG) deviating from normal and assessed as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 millimetres of mercury (mmHg), diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 50 to 90 beats per minute (bpm)
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance, in particular, hepatic parameters (alanine aminotransferase (ALT), aspartate aminotransferase (AST), total bilirubin) or renal parameters (creatinine) exceeding the upper limit of normal (ULN) after repeated measurements
* Any evidence of a concomitant disease assessed as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Cholecystectomy or other surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy or simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures/ convulsions or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or unexplained blackouts

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2021-09-03 (Actual); Primary Completion 2024-07-04 (Actual); Study Completion 2024-07-04 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects with drug-related adverse events | Up to Day 27

SECONDARY OUTCOMES:
Area under the concentration-time curve of the analyte in plasma over a uniform dosing interval of 24 h after administration of the first dose (AUC0-24) | At Day 1
  After the first dose
Maximum measured concentration of the analyte in plasma after the first dose (Cmax) | At Day 1
  After the first dose
Area under the concentration-time curve of the analyte in plasma at steady state over a uniform dosing interval τ (AUCτ,ss) | Up to Day 17
  After the last dose
Maximum measured concentration of the analyte in plasma at steady state over a uniform dosing interval τ (Cmax,ss) | Up to Day 17
  After the last dose
Minimum concentration of the analyte in plasma at steady state over a uniform dosing interval τ (Cmin,ss) | Up to Day 17
  After the last dose
Accumulation ratio based on Cmax,ss (RA,Cmax) | Up to Day 17
  After the last dose
Accumulation ratio based on AUC0-τ (RA,AUC) | Up to Day 17
  After the last dose

CONTACTS AND LOCATIONS:
Locations (1):
- Charité - Universitätsmedizin Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions:
  1. studies in products where Boehringer Ingelheim is not the license holder;
  2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials;
  3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com